CLINICAL TRIAL: NCT02914327
Title: A Phase 1, Open-label Study of SNX-5422 and Ibrutinib in Chronic Lymphocytic Leukemia Subjects With a Mutation in Bruton's Tyrosine Kinase
Brief Title: Safety and Activity of SNX-5422 Plus Ibrutinib in CLL
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Esanex Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNX-5422-CLN1-011
Record Dates: First submitted 2016-09-20; First posted 2016-09-26 (Estimated); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Cancer
Keywords: CLL; Leukemia, Chronic Lymphocytic; Hsp90; BTK; Ibrutinib
MeSH Terms: conditions — Neoplasms; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — SNX-5422; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SNX-5422 plus ibrutinib (Experimental): Open-label administration of SNX-5422 capsules dosed in the morning once every other day for 21 days (11 doses) followed by a 7 day drug free period and daily with the established ibrutinib dose for 28 days of a 28-days cycle. Subjects will repeat the 28-day schedule until the cancer progresses or the subject is unable to tolerate the therapy
  Interventions: Drug: SNX-5422 plus ibrutinib

INTERVENTIONS:
Drug: SNX-5422 plus ibrutinib — SNX-5422 capsule(s) dosed every other day for 21 days out of a 28-day treatment cycle to a total dose of 56 mg/m2 SNX-5422. Subjects will self-administer daily oral ibrutinib in the afternoon at least 8 hours apart from SNX-5422 for 28 days of each cycle.
  Other Names: Imbruvica

SUMMARY:
SNX-5422 is a prodrug of SNX-2112, a potent, highly selective, small molecule inhibitor of the molecular chaperone heat shock protein 90 (HSP90). Hsp90 inhibitors may overcome ibrutinib resistance in Mantle cell lymphomas and this study will investigate whether the addition of SNX-5422 to an established dose of ibrutinib will result in the removal of mutated BTK from blood mononuclear cells and/or prevents or delays disease progression of subjects with CLL

DETAILED DESCRIPTION:
Chronic lymphocytic leukemia (CLL) is the most prevalent leukemia in adults and is not considered curable outside of allogeneic stem cell transplantation.

BTK is a critical kinase in the B cell receptor signaling pathway. This pathway is amplified in CLL and results in amplification of proliferation and anti-apoptotic signals. By inhibiting BTK, ibrutinib eliminates the activation of these pro-survival pathways and microenvironment survival signals. While response to ibrutinib has been high with therapy well-tolerated overall, some patients have relapsed while others have been taken off therapy for toxicity or other reasons. Relapse in CLL can be mediated by at least two separate mechanisms. One is by mutations in BTK, which both decrease ibrutinib's affinity for BTK, and also changes the binding from irreversible to reversible. This is a proof of concept study to investigate whether the addition of SNX-5422 to an established dose of ibrutinib will reduce mutated BTK from CLL cells and/or prevents or delays disease progression of subjects with CLL.

This is an open-label study of SNX-5422 combined with ibrutinib. In each 28 day cycle, SNX-5422 will be dosed in the morning once every other day for 21 days, followed by a 7-day drug-free period. Subjects will continue to receive daily oral ibrutinib at their established dose level in the afternoon every day for 28 days. cycle

ELIGIBILITY:
Inclusion Criteria:

* Males or non-pregnant, non-breastfeeding females 18 years-of-age or older
* A diagnosis of CLL as defined by IWCLL 2008 criteria and currently on treatment with ibrutinib without evidence of disease progression.
* No more than 4 prior lines of anti leukemia therapy (not including ibrutinib)
* Presence of mutated BTK in ≥ 4% of peripheral blood or bone marrow CLL cells, or ≥1% and rising on two separate measurements obtained at least 28 days apart.
* Life expectancy of at least 9 months
* Karnofsky performance score 70
* Adequate baseline laboratory assessments
* Signed informed consent form
* Recovered from toxicities of previous anticancer therapy to CTCAE Grade ≤ 1 with the exception of alopecia
* Subjects with reproductive capability must agree to practice adequate contraception methods.

Exclusion Criteria:

* Subjects experiencing toxicity with ibrutinib
* Prior treatment with any Hsp90 inhibitor.
* Major surgery or significant traumatic injury within 4 weeks of starting study treatment.
* Conventional chemotherapy or radiation within 4 weeks.
* The need for treatment with medications with clinically-relevant metabolism by the cytochrome P450 (CYP) 3A4 isoenzyme within 3 hours before or after administration of SNX-5422
* Screening ECG QTc interval 470 msec for females, 450 msec for males.
* At increased risk for developing prolonged QT interval unless corrected to within normal limits prior to first dose of SNX-5422
* Patients with chronic diarrhea or with Grade 2 or greater diarrhea despite appropriate medical management.
* Gastrointestinal diseases or conditions that could affect drug absorption
* Gastrointestinal diseases that could alter the assessment of safety, including irritable bowel syndrome, ulcerative colitis, Crohn's disease, or hemorrhagic coloproctitis.
* History of documented adrenal dysfunction not due to malignancy.
* History of chronic liver disease.
* Active hepatitis A or B.
* Current alcohol dependence or drug abuse.
* Use of an investigational treatment (except for ibrutinib) from 30 days prior to the first dose
* Glaucoma, retinitis pigmentosa, macular degeneration, or any retinal changes detected by ophthalmological examination that are considered clinically important by examiner.
* Psychological or social reasons that would hinder or prevent compliance with the requirements of the protocol or compromise the informed consent process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of the combination of SNX-5422 and ibrutinib | Every 12 weeks up to 52 weeks
  Change in percent of mutated BTK in CLL cells

SECONDARY OUTCOMES:
Number of subjects reporting adverse events | Day 28 of each 4 week cycle from randomization up to 52 weeks
  Frequency and severity of adverse events
Time to disease progression | Up to 52 weeks
  Elapsed time for each subject from randomization to relapse of disease up to 52 weeks
Clinical Laboratory testing | Day 28 of each 4 week cycle from randomization up to 52 weeks
  Absolute values and changes from baseline for each subject using standard clinical chemistry, hematology and urinalysis parameters
Electrocardiogram | Pre-dose on Day 1 of each 4 week cycle from randomization up to 52 weeks
  Digital 12-lead ECG using standard recording methods at trough drug levels. All ECG recordings will be analyzed for PR, RR, QT intervals, and for morphology.

CONTACTS AND LOCATIONS:
Locations (1):
- Wexner Medical Center, Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No